CLINICAL TRIAL: NCT03836651
Title: A Dietary Intervention to Reduce Inflammation and Oxidative Stress in Persons With Metabolic Syndrome
Brief Title: Dietary Intervention in Persons With Metabolic Syndrome
Acronym: MetLDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martha Biddle (Other)
Responsible Party: Sponsor-Investigator, Martha Biddle, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 45582
Record Dates: First submitted 2019-01-14; First posted 2019-02-11 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Metabolic Syndrome
Keywords: oxidative stress; metabolic syndrome; inflammation
MeSH Terms: conditions — Metabolic Syndrome; Inflammation | interventions — Fruit and Vegetable Juices; Control Groups

STUDY DESIGN:
Intervention Model Description: The design is that of a two-group randomized controlled intervention study. Subjects (N=100) will be randomized to 1 of 2 groups (intervention group or usual care/control group). Subjects will be recruited from outpatient cardiology clinics. The intervention group will be given one 11.5 ounce can of V8® 100% vegetable juice to drink each day for 30 days in addition to their normal diet. The usual care group will continue to consume their normal diet. Data collection for both groups will occur at baseline, and at one-month post-baseline. Data will include sociodemographic and clinical information, 24-hr dietary recalls, carotenoid levels and biomarkers of inflammation and oxidative stress.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Following completion of baseline data collection, participants will be randomized to one of two groups. The research assistant will open a pre-assigned envelope in which group assignment was determined by a random number/block generator. The intervention is designed to complement guideline directed medical management. Therefore, both the intervention and control group will continue to be medically managed by their health care provider as usual. In order to avoid introducing the confound of extra attention paid to the intervention group, the control group will have the same visit and call schedule as the intervention group.
  Interventions: Other: Control group
- Intervention Group (Experimental): Following completion of baseline data collection, participants will be randomized to one of two groups. Participants assigned to the intervention group will receive dietary antioxidants as V8® Low Sodium 100% vegetable juice.
  Interventions: Other: Dietary Antioxidant (V8® Low Sodium 100% vegetable juice)

INTERVENTIONS:
Other: Dietary Antioxidant (V8® Low Sodium 100% vegetable juice) — Following completion of baseline data collection, participants will be randomized to one of two groups. Participants randomized to the intervention group will receive a month's supply of the V8® 100% Low-Sodium Vegetable juice as the dietary antioxidant intervention. Participants will be asked to drink one V8® juice each day for 30 days. Each V8® juice can is 11.5 ounces and can be consumed in divided amounts or all at once. The average daily intake of lycopene is estimated to be 5mg, one can of V8 juice provides 24 mg of lycopene. Thirty days duration for the intervention of V8® juice is based on previous data that indicates plasma antioxidant concentrations rise significantly within a two-week period and a plateau effect is reached within 4 weeks.
  Arms: Intervention Group
Other: Control group — The control group will continue to be medically managed by their health care provider as usual. The control group will have the same visit and call schedule as the intervention group.
  Arms: Control Group

SUMMARY:
Individuals diagnosed with metabolic syndrome are at a two-fold risk for developing cardiovascular disease. The investigators must identify strategies that can abort the development of cardiovascular disease. Inflammation and oxidative stress responsible for the pathogenesis of metabolic syndrome and CVD can be influenced by dietary changes. Strategic and novel interventions that include changing dietary patterns to include more antioxidant rich fruit and vegetables are pragmatic for primary prevention of CVD. Antioxidant rich fruits and vegetables, especially those with carotenoids (lycopene, lutein, zeaxanthin, alpha-carotene, and beta-carotene) have been efficacious in reducing the risk of CVD by decreasing inflammation and oxidative stress. The purpose of this study is to test the effect of a dietary antioxidant intervention on biomarkers of inflammation and oxidative stress in persons diagnosed with metabolic syndrome. The sample will be randomized into one of two groups. Group one (intervention) will drink an 11.5 ounce serving of V8 100% vegetable juice once per day for 30 days. The second group (control) will continue to consume their normal diet. We will measure biomarkers of inflammation (C-reactive protein) and oxidative stress (malondialdehyde) in the two groups at baseline and the end of the 30-day intervention.

DETAILED DESCRIPTION:
SPECIFIC AIMS An estimated 47 million Americans have been diagnosed with metabolic syndrome. Glucose intolerance, abdominal obesity, hypertension and abnormal lipid profile are the identified traits of metabolic syndrome. Metabolic syndrome is a grouping of conditions that collectively are associated with a two-fold risk of cardiovascular disease (CVD). Inflammation and oxidative stress are contributing factors for the development of atherosclerotic plaque in CVD and are the initial pathological responses for each of the abnormal conditions associated with metabolic syndrome. Consequently, reducing inflammation and oxidative stress are considered appropriate targets for interventions designed for primary prevention of CVD and metabolic syndrome. Primary prevention is the fundamental strategy to reduce cardiovascular mortality. Given the high mortality rate associated with CVD and its vast impact on healthcare expenditures, it is imperative that the investigators develop novel interventions for primary prevention of CVD in persons with metabolic syndrome.

Interventions designed to address primary prevention are considered to be the most effective and logical strategy to improve health before the devastating burden of CVD becomes evident. There is an arsenal of CVD treatment modalities available today with many pharmacologic interventions, however, these come at an enormous cost to individuals and to our healthcare system. To address a gap in the treatment of CVD, nonpharmacologic interventions provide an alternative strategy without expense or undesirable adverse side effects. Simple, inexpensive dietary interventions can have a significant impact on an individual's health and are often overlooked by mainstream healthcare providers because of their simplicity. The impact of increasing fruit and vegetables, which are loaded with antioxidants, into a dietary pattern has consistently been supported in research and is recommended in all primary prevention guidelines. Yet, nine out of ten Americans get less than the recommended amounts of fruits and vegetables in their diet.

The purpose of this study is to test the effect of a dietary antioxidant intervention on inflammation and oxidative stress in individuals with metabolic syndrome. The study has the potential to reduce the incidence of cardiovascular disease. This proposal will address a major goal of Healthy People 2020: Improving cardiovascular health through prevention, detection, and treatment, specifically addressing primary prevention of CVD in individuals with metabolic syndrome.

Specific Aim #1: To test the effect of a dietary antioxidant intervention on biomarkers of inflammation and oxidative stress in individuals who have metabolic syndrome.

Hypothesis #1: Compared to a usual care control group and to their own baseline, individuals randomized to a dietary antioxidant intervention (30-day intake of V8® 100% Low-Sodium Vegetable juice) group will have lower levels of C-reactive protein (CRP) and malondialdehyde (MDA) at one month from baseline. CRP is a biomarker of inflammation and is an independent predictor of cardiovascular disease. MDA is the most prevalent byproduct of lipid peroxidation during oxidative stress and is considered an excellent measurement for use in clinical trials to evaluate oxidative stress.

ELIGIBILITY:
Inclusion Criteria: Subjects will be individuals who have a diagnosis of metabolic syndrome without overt CVD as defined by the National Cholesterol Education Program (NCEP) as evidenced by having at least 3 of the 5 following conditions:

1. Hypertension defined as SBP >130mmHg and diastolic >85mmHg
2. Abdominal obesity with a waist circumference greater than 88cm in women and greater than 102 cm in men
3. Triglycerides level greater than 150mg/dL
4. HDL levels less than 50mg/dL in women and less than 40mg/dL in men
5. Fasting glucose level greater than 100mg/dL Additional inclusion criteria include the ability to read and speak English, and have no cognitive impairment that precludes giving informed consent or ability to follow protocol instructions.

   -

   Exclusion Criteria: Subjects will be excluded from the study if they: a) are less than 21 years of age; b) have a terminal illness; c) have impaired cognition; d) have a strong dislike, or have a potential food-drug interaction to V8® Low Sodium 100% vegetable juice; or e) co-existing illness documented in the medical record or self-reported associated with systemic inflammation (e.g. rheumatoid arthritis, acute systemic infection).

   -

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Change in plasma C-reactive Protein (CRP) from baseline to one month. | Baseline and one month
  Plasma will be collected at baseline and one month (up to 30 days) later for analysis of CRP. Data will be presented as the change over time between groups.

SECONDARY OUTCOMES:
Change in plasma Malondialdehyde (MDA) from baseline to one month. | Baseline and one month
  Plasma will be collected at baseline and one month (up to 30 days) later for analysis of MDA. Data will be presented as the change over time between groups.

OTHER OUTCOMES:
Diet quality: Healthy Eating Index score | up to 30 days
  The 24-hour dietary recall will be collected at baseline, two weeks into the study and one month (about 30 days) after study initiation by phone call.
  Each food recall time point will be analyzed using the Nutrition Data System for Research (NDSR) software program and used to measure diet quality. The food quality assessment will be presented as the change in dietary quality (Healthy Eating Index score) over time between groups.
Change in skin tissue Carotenoid levels at baseline and 1 month. | Baseline and one month
  Skin carotenoid levels will be measured at baseline and 1 month (up to 30 days) using reflection spectroscopy approach (Veggie Meter) to determine adherence to the dietary intervention. Carotenoid levels will be presented as the change over time between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Biddle, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No